# Study Protocol

# Naloxone for Optimizing Hypoxemia of Lung Donors (NO-HOLDS)

### NCT02581111

Date: August 14, 2015

#### **Project Goals**

- 1. Evaluate whether naloxone can improve oxygenation / reverse hypoxemia in lung-eligible braindead (BD) organ donors
- 2. Demonstrate feasibility of prospective multi-OPO clinical trials as part of the ODRC

### Study Population (determined at initiation of OPO management)

- 1. Lung-eligible BD donors (age 13-70, no established severe lung disease e.g. COPD)
- 2. Arterial hypoxemia (P:F ratio < 300 on first ABG after initial OPO stabilization)

#### Study Protocol

- 1. All OPO-specific donor protocols (incl. lung optimization) should be followed
  - a. Does not require any other change to practice or donor management
- 2. Randomization occurs for eligible donors after initial ABG (stratified by center)
- 3. Naloxone 8 mg IV (or saline) given once
  - a. Co-administered with a neuromuscular blocking agent (NMB)
  - b. Blinding of drug vs. placebo done at each OPO with sequential unmarked syringes (prefilled with naloxone or saline and numbered with central code)

#### **Outcome Measures**

- 1. Change in P:F ratio to final ABG ABG obtained on 100% FiO2, PEEP 5
- 2. Change in P:F ratio to early ABG
- 3. Lungs recovered / transplanted (if not reason, e.g. hypoxemia vs. COPD, other RO)

SRTR variables for O:E calculation (incl. age, race, ABO, smoker)

- Most of this could be abstracted post-hoc from OPO database
- Only study registration (with UNOS & OPO ID) entered into study-specific on-line database with syringe # and ABG PO<sub>2</sub> values (<u>redcap.wustl.edu</u>)